CLINICAL TRIAL: NCT06495359
Title: Effect of Immunization Education Program on Parental Vaccine Hesitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aslı Akdeniz Kudubeş, ASSOCIATE PROFESSOR, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: aslıkudubes
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Nurse's Role
Keywords: Immunization; Parents; Education

STUDY DESIGN:
Intervention Model Description: A parallel group (experiment-control) randomized controlled design, which is one of the experimental methods
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Researchers will administer the immunization education program to parents.
  Interventions: Other: immunization education program
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: immunization education program — The content of the immunization education program for parents was created by researchers based on the literature. Expert opinions will be obtained from 7 people who are experts in the fields of child health and disease nursing and public health nursing for the training program. The training program consists of 30 minutes. The education program will be delivered to parents in the form of a 30-minute training session using the face-to-face education model. Interactive education methods that enable parents' participation will be used.
  Arms: Experimental group

SUMMARY:
Not administering vaccines due to vaccine hesitancy is both a potential public health problem and a difficult and risky situation for healthcare professionals. Health sector workers play a very important role in vaccinating families. As public awareness increases, interest in these vaccines is likely to increase. Made works; It shows that healthcare professionals and physicians establishing trust and communicating effectively with vaccine recipients and parents is one of the most effective ways to eliminate vaccine hesitations. They stated that in order for childhood vaccines to be administered at a high rate, effective communication should first be established with parents. This project aimed to determine the effect of the immunization education program on parents' vaccine hesitancy. The project is designed as a randomized controlled study and will consist of experimental and control groups. An education program regarding immunization will be applied to the parents in the experimental group. The originality of this project is the evaluation of the effect of the immunization education program applied to parents whose children are hospitalized on vaccine hesitancy. Although studies on vaccine hesitancy in parents have increased in recent years, most of them consist of descriptive studies aimed at determining the level of vaccine hesitancy and affecting factors. No intervention studies on the effect of immunization education in parents on vaccine hesitancy have been found.

DETAILED DESCRIPTION:
The aim of the research will be carried out using a parallel group (experiment-control) randomized controlled design, which is one of the experimental methods, to determine the effect of the immunization education program on parents' vaccine hesitancy.

Goals:

* To examine the effect of the immunization education program on parents' vaccine hesitancy,
* To compare the average scores of the vaccine hesitancy scale between the parents in the experimental group and the control group in the project.

ELIGIBILITY:
Inclusion Criteria:

* Having a child between the ages of 0-6,
* admitted to the pediatric ward,
* who have not previously received training on immunization
* Parents who volunteered to participate in the study

Exclusion Criteria:

* illiterate
* parents with mental retardation, vision and hearing impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Parental Vaccination Hesitancy Scale mean score | up to 10 months
  The effect of the applied education on the mean score of the Parental Vaccination Hesitancy Scale will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: AKDENİZ KUDUBEŞ, Study Director — BİLECİK ŞEYH EDEBALİ UNIVERSITY
Locations (1):
- Asli Akdeniz Kudubeş, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No